CLINICAL TRIAL: NCT02165813
Title: A Randomised, Placebo-controlled Trial of Oral Nitazoxanide for the Empiric Treatment of Acute Gastroenteritis Among Australian Indigenous Children
Brief Title: Oral Nitazoxanide in Acute Gastroenteritis in Australian Indigenous Children
Acronym: NICEGUT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Continuation of enrolment was deemed not feasible due to very small eligibility numbers and funding exhausted.
Sponsor: Telethon Kids Institute (Other)
Collaborators: The University of Western Australia (Other); Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NICEGUT
Record Dates: First submitted 2014-06-09; First posted 2014-06-18 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Bayesian piecewise survival analysis
Who Masked: Participant, Care Provider, Investigator
Masking Description: Matched placebo formulation
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitazoxanide (Active Comparator): oral nitazoxanide suspension twice daily for 3 days
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): oral placebo suspension twice daily for 3 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide is a synthetic drug of the nitrothiazolide class. The main metabolite of NTZ is tizoxanide. The active ingredient is Nitazoxanide (2-acetyloxy-N(5-nitro-2-thiazolyl)benzamide), a synthetic agent for oral administration, at a concentration of 100 mg/5 ml.
  Other Names: Alinia
  Arms: Nitazoxanide
Drug: placebo — An oral suspension is supplied as a pink coloured powder formulation (sugar) that is reconstituted with 48 mL water prior to use to a final volume of 60 mls.
  Arms: Placebo

SUMMARY:
This is a multi-centre (RDH and ASH), phase IV, double-blind, randomised, placebo-controlled Bayesian adaptive trial of oral NTZ for the treatment of acute gastroenteritis requiring admission to hospital. A maximum of 300 children aged between three months and less than five years of age will be enrolled. Study participation is from the point of enrolment until 60 days after enrolment. Enrolment will occur within 48 hours of admission to hospital. Enrolled participants will be randomised 1:1 to Nitazoxanide (NTZ) or placebo. Other treatment and management will be as per the standard of care described in the admitting hospital's guidelines and will be ultimately the decision and responsibility of the named medical consultant. Stool samples will be collected at the point of admission. Solicitation of symptoms will be by review of routinely collected medical data recorded in the participant's medical record, and will be supplemented by completion of study specific diary cards after discharge (for the first 210 enrolments). Attempts will be made to contact participants at day 7 after enrolment (by telephone if already discharged) to ascertain symptoms occurring in the intervening period. At days 30 and 60 (for first 210 enrolments ) and Day 60 (for enrolment #211 onwards) after enrolment a clinical record review will be conducted for all participants to ascertain health care attendances following discharge.

DETAILED DESCRIPTION:
This is a multi-centre (RDH and ASH), phase IV, double-blind, randomised, placebo-controlled Bayesian adaptive trial of oral NTZ for the treatment of acute gastroenteritis requiring admission to hospital. A maximum of 300 children aged between three months and less than five years of age will be enrolled. Study participation is from the point of enrolment until 60 days after enrolment. Enrolment will occur within 48 hours of admission to hospital. Enrolled participants will be randomised 1:1 to Nitazoxanide (NTZ) or placebo. Other treatment and management will be as per the standard of care described in the admitting hospital's guidelines and will be ultimately the decision and responsibility of the named medical consultant. Stool samples will be collected at the point of admission. Solicitation of symptoms will be by review of routinely collected medical data recorded in the participant's medical record, and will be supplemented by completion of study specific diary cards until discharge (for the first 210 enrolments). Attempts will be made to contact participants at day 7 after enrolment (by telephone if already discharged) to ascertain symptoms occurring in the intervening period. At days 30 and 60 (for first 210 enrolments ) and Day 60 (for enrolment #211 onwards) after enrolment a clinical record review will be conducted for all participants to ascertain health care attendances following discharge.

The sample size for the study is a maximum of 300 children, randomised on a 1:1 basis to the two study treatment groups. The trial will stop recruiting when pre-specified decision criteria are met based on treatment superiority or trial futility or when 300 children have been enrolled. Based on previously published data it is hypothesised that NTZ treatment will result in a decrease in the median duration of medically significant illness by 1 day. A decrease of one day is considered to be the minimum useful decrease of relevance to the study setting. It is anticipated that there will be minimal lost to follow-up as the primary endpoint will be available for the majority of participants in each arm due to the short interval between enrolment and meeting the criteria for the primary endpoint.

The trial will be conducted as a fixed allocation Bayesian adaptive randomised controlled trial. This statistical methods in the protocol are written to be practical and accessible to individuals with an understanding of common clinical trial designs and classical frequentist analytical methods but without training in Bayesian statistics. A formal description of the interim Bayesian data analysis fundamental to this design, which assumes substantial familiarity with Bayesian calculation of posterior distributions conditioned on observed data, is documented in the Statistical Analysis Plan. There is overlap between the protocol and statistical analysis plan so that each may serve an appropriate audience as a standalone description of the statistical methods. Briefly, within the Bayesian framework, the intervention arms are evaluated and sequential Bayesian statistical analyses are used over time to incorporate new trial outcome information to determine if a treatment is superior, inferior, or equivalent, with respect to the primary end-point. Every child will be randomly assigned in a ratio 1:1 to placebo or nitazoxanide. Children will be classified by membership in different strata, where membership will be defined by age and geographical region. Whenever an interim analysis reports superiority, inferiority, or equivalence with respect to the primary end-point this is termed a Statistical Trigger. At any given interim analysis, a Statistical Trigger may be reached for all children or for one or more strata.

ELIGIBILITY:
Inclusion Criteria:

1. Infant /child between =>3 months and <5 years of age
2. Infant/ child identified as Indigenous by the legally responsible care-giver
3. Infant /child has been/will be admitted to hospital for acute infectious gastroenteritis (in the opinion of the admitted doctor and/or study doctor/nurse )
4. The legally responsible care-giver is willing for their infant/ child to participate in the study and who would be expected to comply with the requirements of the protocol, including being able and willing to be contacted by telephone after discharge where necessary
5. The legally responsible care-giver is willing to allow other parties involved in the treatment of his or her child (including the general practitioner, paediatrician, hospital medical and nursing staff, community clinic staff) to be notified of participation in the trial
6. The legally responsible care-giver is willing to allow to allow the study team to obtain a vaccination history from Australian Childhood Immunisation Register (ACIR) and/or local provider
7. The legally responsible care-giver is willing to allow the study team to obtain an interim medical history from the participant's electronic medical records and/or from the participant's general practitioner for the period from enrolment to study day 60
8. Informed consent for the infant's/child's participation in the study has been given by the legally responsible care-giver

Exclusion Criteria:

1. Admitted for =>48 hours at the point of enrolment
2. Duration of symptoms of greater than 14 days without apparent worsening of symptoms consistent with an acute pathology
3. Presence of grossly bloody diarrhoea
4. Clinical suspicion of non-infectious cause (e.g. diagnosed with a pre-existing medical condition predisposing to non-infectious diarrhoea, for example inflammatory bowel disease) except for environmental enteropathy)
5. Contraindication to the study drug or placebo (e.g. allergy)
6. Diagnosis of infection with an enteric pathogen where anti-microbial treatment with an alternative antimicrobial is the standard of care (e.g. Shigella sp.)
7. Inability to tolerate either the oral or nasogastric route (e.g. ileus)
8. Clinical suspicion of intestinal obstruction including bilious vomiting
9. Confirmed or suspected immunosuppressive or immunodeficient conditions, including human immunodeficiency virus (HIV) infection.
10. Receipt of more than 2 weeks of immuno-suppressants or immune modifying drugs, (e.g. prednisolone >0.5 mg/kg/day)
11. Receipt of investigational drug/vaccine, other than the drugs used in the study, within 30 days prior to receiving the first dose of NTZ or their planned use during the study period, until 1 month after the administration of the final dose of NTZ
12. Previously enrolled in the trial

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Time of significant illness | Between randomisation and hospital discharge (expected to be within 7 days)
  The time period of significant illness (defined as the period for which hospitalisation is required for medical reasons) for participants in each study treatment group.

SECONDARY OUTCOMES:
Time to hospital discharge | Between randomisation and hospital discharge (expected to be within 7 days)
  The time period between enrolment and actual discharge from hospital

OTHER OUTCOMES:
Symptom frequency (vomiting, diarrhoea, generally unwell) | On each of study days 0-7
  The proportion of participants experiencing each solicited symptom (vomiting, diarrhoea, generally unwell) on each of study days 0-7
Dehydration frequency and severity | On each of study days 0-7
  The proportion of participants in whom dehydration is present and the severity of dehydration, where present, on each study day using a protocol-specific dehydration score from 0 (not dehydrated) to 3 (severely dehydrated)
Time of intravenous, intraosseous or nasogastric rehydration | 7 days post randomisation
  The time interval between either starting intravenous, intraosseous or nasogastric rehydration or enrolment (whichever is the later), and ceasing rehydration or discharge for the first 210 participants.
Severity score for each adverse event | 0-60 days post randomisation
  The maximum daily severity score for each adverse event , where experienced. Will be assessed using a protocol-specific grading system from 0 (normal) to 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Tom Snelling, Principal Investigator — Sydney University
Locations (2):
- Australia (2):
  - Alice Springs Hospital, Alice Springs, Northern Territory
  - Royal Darwin Hospital, Darwin, Northern Territory

REFERENCES:
- [Background] Waddington CS, McLeod C, Morris P, Bowen A, Naunton M, Carapetis J, Grimwood K, Robins-Browne R, Kirkwood CD, Baird R, Green D, Andrews R, Fearon D, Francis J, Marsh JA, Snelling T. The NICE-GUT trial protocol: a randomised, placebo controlled trial of oral nitazoxanide for the empiric treatment of acute gastroenteritis among Australian Aboriginal children. BMJ Open. 2018 Feb 1;8(2):e019632. doi: 10.1136/bmjopen-2017-019632. PMID 29391385
- See also: Related Info — https://bmjopen.bmj.com/content/8/2/e019632